CLINICAL TRIAL: NCT05448534
Title: Electroencephalographic Patterns of Septic Patients and Its Correlation With Cognitive Outcomes
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, ICU Coordinator, Hospital Sao Domingos
Other Study IDs: 54
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Sepsis
Keywords: Eletroencephalography; Sepsis; Septic shock; Critical care; cognitive dysfunction; Montreal cognitive assessment
MeSH Terms: conditions — Sepsis; Shock, Septic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Eletroencephalography — We used Sinek and Young Scale to classify electroencephalographic patterns and cognitive outcome with MOCA score.
  Other Names: Montreal Cognitive Assessment (MoCA); Sinek and young scales

SUMMARY:
The investigators evaluated the electroencephalographic pattern by the Sinek and Young scales during ICU stay and its correlation with cognitive impairment determined by the Montreal Cognitive Assessment (MOCA) in septic patients after 3 months of ICU discharge..

DETAILED DESCRIPTION:
The investigators prospectively evaluate patients with sepsis and septic shock expected to stay in the intensive care unit (ICU) for at least 4 days. We used Sinek and Young scales to classify electroencephalographic patterns during ICU stay (in the first 24 hours after admission and in the third ICU day) and correlate with cognitive outcome evaluated with MOCA score 3 months after ICU discharge. The investigators evaluate as primary outcome the association between electroencephalographic abnormalities and cognitive dysfunction measured by the Montreal Cognitive Assessment (MoCA) 3 months after ICU discharge and secondary outcomes as association between electroencephalographic patterns and 28 days mortality, Quality of Life (SF-36) after 3 months of discharge, ventilator free days, vasoactive drug free days and Glasgow outcome scale.

ELIGIBILITY:
Inclusion Criteria:

Included were patients aged above 18 years, who were expected to stay in the ICU for at least 4 days, between November 2021 and November 2022.

-

Exclusion Criteria:

* CNS infections,
* Structural abnormalities of the CNS, known
* Liver or uremic encephalopathy,
* Advanced dementia (Mini mental < 9),
* Psychiatric disorder
* Epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill patients with sepsis and septic shock expected to stay in the intensive care unit (ICU) for at least 4 days admitted to 3 medical ICUs and 2 surgical ICUs of a tertiary hospital in Brazil.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Electroencephalographic patterns | 3 months after hospital discharge
  Electroencephalographic patterns determined by Sinek and Young scales. The Synek outcome Scale ranges from normal (alpha dominant rhythm) to suppression (worst outcome). The scale assesses the outcome of patients with sepsis.
  Young's Scale Electroencephalographic classification of coma assesses outcome of patients with sepsis Outcome varies from normal (Delta/Theta Rhythm > 50% of record). worst result Suppression The two scales are complementary.
Cognitive evaluation | 3 months after hospital discharge
  Cognitive dysfunction measured by Montreal Cognitive Assessment (MoCA)

SECONDARY OUTCOMES:
electroencephalographic patterns and 28 days mortality . | 28 days
  Electroencephalographic patterns determined by Sinel and Young scales and 28 days .mortality. The Synek outcome Scale ranges from normal (alpha dominant rhythm) to suppression (worst outcome). The scale assesses the outcome of patients with sepsis.
  Young's Scale Electroencephalographic classification of coma assesses outcome of patients with sepsis Outcome varies from normal (Delta/Theta Rhythm > 50% of record). worst result Suppression The two scales are complementary.
Quality of Life (SF-36) after 3 months of discharge | 3 months after hospital discharge
  Quality of life determined through Short-Form Health Survey (SF-36). Scores range from 0 to 100, 0 indicating the less favorable health status and 100 the most favorable one.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE AZEVEDO, MD, PhD, Study Director — Hospital Sao Domingos
Locations (1):
- Icu Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Azabou E, Magalhaes E, Braconnier A, Yahiaoui L, Moneger G, Heming N, Annane D, Mantz J, Chretien F, Durand MC, Lofaso F, Porcher R, Sharshar T; Groupe d'Explorations Neurologiques en Reanimation (GENER). Early Standard Electroencephalogram Abnormalities Predict Mortality in Septic Intensive Care Unit Patients. PLoS One. 2015 Oct 8;10(10):e0139969. doi: 10.1371/journal.pone.0139969. eCollection 2015. PMID 26447697
- [Result] Eidelman LA, Putterman D, Putterman C, Sprung CL. The spectrum of septic encephalopathy. Definitions, etiologies, and mortalities. JAMA. 1996 Feb 14;275(6):470-3. PMID 8627969
- [Result] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Result] Oddo M, Carrera E, Claassen J, Mayer SA, Hirsch LJ. Continuous electroencephalography in the medical intensive care unit. Crit Care Med. 2009 Jun;37(6):2051-6. doi: 10.1097/CCM.0b013e3181a00604. PMID 19384197
- [Result] Young GB, Bolton CF, Archibald YM, Austin TW, Wells GA. The electroencephalogram in sepsis-associated encephalopathy. J Clin Neurophysiol. 1992 Jan;9(1):145-52. doi: 10.1097/00004691-199201000-00016. PMID 1552002
- [Result] Hosokawa K, Gaspard N, Su F, Oddo M, Vincent JL, Taccone FS. Clinical neurophysiological assessment of sepsis-associated brain dysfunction: a systematic review. Crit Care. 2014 Dec 8;18(6):674. doi: 10.1186/s13054-014-0674-y. PMID 25482125